CLINICAL TRIAL: NCT06734715
Title: Oxy-PICU Neurodevelopmental Follow-up Study
Acronym: Oxy-PICU ND
Status: Not yet recruiting | Type: Observational
Sponsor: Intensive Care National Audit & Research Centre (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Oxy-PICU ND v1.0; NIHR206910 (Other Grant/Funding Number: National Institute for Health and Care Research (NIHR) Research for Patient Benefit (RfPB))
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Intensive Care Pediatric
Keywords: Neurodevelopment; Paediatric critical care; Oxygen

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conservative oxygenation: Patients that have previously received treatment in paediatric intensive care with conservative oxygenation
  Interventions: Other: Conservative oxygenation
- Liberal oxygenation: Patients that have previously received treatment in paediatric intensive care with liberal oxygenation
  Interventions: Other: Liberal oxygenation

INTERVENTIONS:
Other: Conservative oxygenation — Patients that were previously randomised to receive conservative oxygenation while in paediatric intensive care
  Groups: Conservative oxygenation
Other: Liberal oxygenation — Patients that were previously randomised to receive conservative oxygenation while in paediatric intensive care
  Groups: Liberal oxygenation

SUMMARY:
Background to the research: Each year around 20,000 children are admitted to paediatric intensive care units (PICUs) in the UK. Of these children, ~75% will receive support from a breathing machine (or ventilator) in combination with additional oxygen. We recently completed the NIHR funded Oxy-PICU randomised clinical trial (RCT) - a study that compares one treatment against another to determine which is best. The Oxy-PICU RCT investigated whether children in PICU who are receiving help from a ventilator with additional oxygen, should have their oxygen levels kept at a lower level or higher level which currently used in the NHS. We found that aiming for lower oxygen levels was better and resulted in a small but significant reduction in the number of days children spent on machines or died at 30 days.

While small, this result would have a large and important impact for patients and their families and may have important cost savings for the NHS. However, while in the short-term targeting lower oxygen levels appears better, the effects on children's longer-term development are unknown. Knowing this is important to fully inform doctors and nurses about the effects of aiming for lower oxygen levels, and help the results of Oxy-PICU be applied throughout the NHS.

Aim of the research: This research aims to complete longer-term follow-up of children included in the Oxy-PICU RCT. We will look at the effect of aiming for lower oxygen levels compared to higher oxygen levels on longer-term developmental milestones.

Research plan: We will invite 1,112 parents of children included in the Oxy-PICU RCT by email and post to take part. We will arrange a telephone interview with the parent(s) who agree to participate. A trained researcher will use standard questionnaires to measure important issues. They'll establish if the children are meeting their developmental milestones and learn about their health related quality of life. After the interview we will provide a report to the parents detailing their child's development. We anticipate 50% of those approached will agree to take part in this study. This will allow us to detect important differences in developmental milestones in children treated with lower oxygen levels.

Patient and public involvement: PPI has been essential throughout Oxy-PICU. Our PPI co-applicant has been involved in Oxy-PICU from the start as a key member of the study team and will continue to help oversee all aspects of this research. We will also appoint a parent advisory group to provide additional PPI input into the study processes.

Knowledge mobilisation: Outputs from the neurodevelopmental follow-up will be specifically targeted to the key stakeholders including patients/parents, clinicians and policy makers. Outputs for patients/parents and the public will be co-produced with our PPI representatives.

DETAILED DESCRIPTION:
Research question: In invasively ventilated critically ill children referred as an emergency for paediatric intensive care receiving supplementary oxygen [Population] what are the effects of a conservative oxygen therapy [Intervention] compared with a liberal oxygen therapy [Comparator] on longer-term neurodevelopmental function [Outcome]?

Background: We recently completed the NIHR funded Oxy-PICU randomised clinical trial (RCT) which compared conservative versus liberal oxygenation targets in emergency admissions to PICU receiving invasive mechanical ventilation. The results showed a small but significant reduction in the number of days spent receiving organ support or death by day 30 with conservative oxygenation. While the effect size, in terms of the primary outcome, may appear small, if true, these results are clinically important to patients/parents and the NHS. While conservative oxygenation appears effective in the short term, questions still remain about the effects of targeting lower oxygen saturations on longer-term neurodevelopmental function, with calls made from PICU clinicians for this to be investigated prior to wider spread adoption of the Oxy-PICU trial results.

Aim: to extend and undertake additional follow-up of children enrolled in the Oxy-PICU RCT, to determine the effects of conservative oxygen therapy on longer-term neurodevelopmental function in critically ill children.

Methods: 1,112 parents of children included in the Oxy-PICU RCT will be invited by email and post to take part in this longer-term follow-up study. After agreeing to participate, we will arrange a telephone interview with the parent(s) consisting of two validated questionnaires: 1. Vineland Behaviour Scales, third edition (VABS-3) and 2. PedsQL™ 4.0 (Pediatric Quality of Life Inventory) which provide a validated proxy for neurodevelopmental functioning and quality of life, respectively. Once the interview has been completed, we will provide a report to the parents detailing their child's development.

Primary outcome: neurodevelopmental function defined as the overall adaptive behaviour VABS-3 score.

Sample size: Anticipating 50% of those approached agreeing to take part in this study, 556 parents completing telephone interviews will provide enough people to detect a clinically important difference in neurological and developmental function in children treated with conservative oxygen saturations compared with higher oxygen saturations.

Timeline: Total duration: 24 months: months 1-3: HRA approval and interview training; months 4-21: patient/parent recruitment and telephone interviews; months 22-24: analysis and dissemination.

Impact and dissemination: This research will have a large and immediate impact on patients, parents/guardians and the NHS. Understanding the neurodevelopmental effects of conservative oxygen therapy is imperative for implementation of the Oxy-PICU results, which has the potential for important clinical benefit for critically ill children and the NHS. We will actively disseminate the results of the Oxy-PICU neurodevelopmental follow-up study with specific outputs targeted at patients and the public, PICU clinicians/researchers and policy makers. Outputs targeting patients and public will be co-designed with PPI representatives.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or caregiver of child included in the Oxy-PICU RCT;
2. Provided consent to be contacted about future research;
3. Living with child; and
4. Child/young person survival status confirmed.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents/caregivers of children enrolled into Oxy-PICU and who provided consent to be contacted about future related research.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental function defined as the overall adaptive behaviour score assessed using the Vineland Adaptive Behaviour Scales, third edition (VABS-3). | 4 years post randomization into the Oxy-PICU RCT (ISRCTN92103439)
  Overall adaptive behaviour score obtained from the Vineland Adaptive Behaviour Scales, third edition (VABS-3) questionnaire.

SECONDARY OUTCOMES:
VABS-3 domain scores | 4 years post randomization into the Oxy-PICU RCT (ISRCTN92103439)
  Individual VABS-3 domain scores (communication, daily living skills, socialisation, motor skills in younger children)
Health related quality of life | 4 years post randomization into the Oxy-PICU RCT (ISRCTN92103439)
  Health related quality of life (HRQoL) measured using the Pediatric Quality of Life Inventory (PedsQL™) 4.0.

IPD SHARING:
Plan to Share IPD: Undecided